Study title: Sub-Ischial Socket for Transfemoral Amputation and Lower Mobility

NCT number: NCT05662982

**Document:** University of Washington and Hanger Clinic ICF - reference group (version 08/31/2023)

# UNIVERSITY OF WASHINGTON AND HANGER CLINIC CONSENT FORM

**Evaluation of the Northwestern University Sub-Ischial Socket for Persons with Transfemoral Amputation and Lower Mobility Levels (reference group)** 

| Stefania Fatone, PhD, BPO(Hons), Professor, UW Rehabilitation Medicine | 206-685-7918 |
|---|---|
| Shane Wurdeman, PhD, Director, Clinical Research, Hanger Clinic | 402-290-8051 |
| Siya Asatkar, BA, Research Assistant, Hanger Clinic | 512-774-7105 |
| Dana Wilkie, Research Coordinator, Rehabilitation Medicine | 206-221-2414 |
| Alexandra Hinson, Research Assistant, Rehabilitation Medicine | 206-221-2414 |

#### Researchers' Statement

We are asking you to be in a research study. This form gives you information to help you decide whether or not to be in the study. Being in the study is voluntary. Please read this carefully. You may ask any questions about the study. Then you can decide whether or not you want to be in the study.

#### **KEY STUDY INFORMATION**

This research study will determine whether a new prosthetic socket design, which is supposed to be more comfortable than current prosthetic socket designs, will help people with amputation wear the socket more and therefore walk more. We are inviting you to take part in the study because you have an above-the-knee amputation and wear a prosthesis. This page is to give you key information to help you decide whether or not to participate. Ask the research team questions. If you have questions later, the contact information for the research investigator in charge of the study is above.

# WHY ARE WE DOING THIS STUDY AND WHAT WILL YOU BE ASKED TO DO IF YOU PARTICIPATE?

We are asking you to participate in this study as a reference subject so we can have comparison data from people who wear prosthesis in the community. As a reference subject we will monitor you in your usual prosthesis for 10 months. This will be done by asking you to complete a total of 8 surveys remotely (online, on paper, or by phone) every 4 to 8 weeks.

# WHY MIGHT YOU NOT WANT TO BE IN THIS STUDY?

It is also possible that being repeatedly asked questions about your everyday life (e.g. symptoms of depression) may be upsetting.

#### WHY MIGHT YOU WANT TO BE IN THIS STUDY?

Collecting data from a reference group of participants will help us assess if the new socket is more comfortable and improves the ability to get around for other people with amputation.

#### DO YOU HAVE TO TAKE PART IN THE STUDY?

If you decide to take part in the study, it should be because you really want to volunteer. If you decide not to take part, you will not lose any services, benefits, or rights you would normally have. You will still receive treatment from your prosthetist. You can choose to withdraw at any time during the study.

# What is the purpose of the study?

The purpose of this research is to determine whether a new prosthetic socket design, which is supposed to be more comfortable than current prosthetic socket designs, will help people like you wear the socket more and therefore walk more. Your role in this study is to provide reference data about what happens over time when the socket remains the same.

# What does my participation in the study involve?

Participation in this study will last about 10 months and involves 8 remote survey assessments.

We will collect basic information about your amputation and your current socket and prothesis from your medical record. You will complete the same survey (either online, on paper, or by telephone) every 4 to 8 weeks for a total of 8 times. The survey includes questions about how your current socket influences your everyday life, including questions about socket comfort, mobility, and balance, as well as questions about your physical and emotional well-being, including symptoms of depression. You may refuse to answer any question. Each survey assessment will take about 30 minutes to complete. Summary of the study sessions:

| Study<br>Session | When | Location | Study Activity | Duration | Payment for completed session |
|---|---|---|---|---|---|
| Sessions<br>1 - 8 | Weeks<br>0, 4, 8, 12, 20,<br>28, 36 & 40 | Home or place convenient for you | 1 survey/<br>session | 30 minutes/<br>session | \$25/session<br>\$50: bonus for<br>completing all<br>sessions |

#### What are the risks?

Being in this study will expose you to some risks:

- It is possible that you may experience fatigue and/or boredom while answering the survey questions.
- There is the risk that being asked questions about your everyday life, such as symptoms of depression and/or mental well-being, may be upsetting.
- It is possible that someone could find out you were in this study and could find out information about you. The researchers have procedures in place to lessen the possibility of this happening.

## Are there alternatives to participating in this study?

You can choose not to be in the study.

## Are there any benefits to participating in this study?

You will not experience any direct benefit from being in the study.

## Who is funding this study?

The University of Washington is receiving financial support from the Department of Defense. Hanger Clinic is receiving financial support for this research from the United States Department of Defense (DOD) under a subcontract from University of Washington.

Consent Form, SI Socket Study, Reference

### How is my information kept confidential?

All the information you provide will be confidential. Your name and other identifying information will be linked to a unique study number. Your study number will not include any information that can identify you. All data we collect from you will be coded with your study number and stored securely. The study team will use REDCap, an online database to collect and store your information. The information in REDCap will include information that will identify you, such as your name and contact information. REDCap is a secure system for data storage used in many research studies. REDCap requires a username and password to log-on and is encrypted. REDCap is stored on a secure server. The study team is able to choose who has access to log-on to REDCap and see your information. Access will only be given to Hanger Clinic and University of Washington study team members. The link between your identifying information and study data will be destroyed after the record retention period required by law.

Government or university staff sometimes review studies such as this one to make sure they are being done safely and legally. If a review of this study takes place, your records may be examined. The reviewers will protect your privacy. The study records will not be used to put you at legal risk of harm.

The U.S. Food and Drug Administration (FDA) reserves the right to review study data that may contain identifying information.

Organizations that may inspect and copy your information include the IRB and other representatives of this institution, the US Department of Defense (DOD), the DOD Human Research Protections Office, the Veterans Administration, and collaborators at Hanger Clinic. By signing this document, you are authorizing this access.

A description of this clinical trial will be available on <a href="http://www.clinicaltrials.gov">http://www.clinicaltrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

If a research staff member finds out you have plans or intent to harm yourself or others, s/he may refer you to or contact an appropriate individual or institution. We will not ask you about child or elder abuse, but if you tell us about child or elder abuse or neglect, we may be required or permitted by law or policy to report to authorities.

You may be withdrawn from the study without your consent if the researchers believe it is in your best interest or if you are not able to fulfill the study requirements.

## Will I be paid for taking part in this study?

If you agree to take part in this research study, we will pay you \$25 per survey assessment for up to 8 assessments. We will pay you a bonus of \$50 at study completion if you complete all 8 survey assessments. If you complete all study sessions, you would receive a total of \$250. You will receive payment via check within 2-4 weeks of each study session. You will only be paid for the study sessions you complete.



# How will my study information be used?

We may publish the results of this research. However, we will keep your name and other identifying information confidential.

The information that we obtain from you for this study might be used for future studies. We may remove anything that might identify you from the study information. If we do so, that information may then be used for future research studies or given to another investigator without getting additional permission from you. It is also possible that in the future we may want to use or share study information that might identify you. If we do, the UW Human Subjects Division will decide if we need to get additional permission from you.

We will not provide you with your individual results from this study.

## Is there anything else I should know about the study?

You may refuse to participate and you are free to withdraw from this study at any time without penalty or loss of benefits to which you are otherwise entitled. If you wish to withdraw, please contact the researcher listed on page 1 of this consent form.

For female participants, because a pregnancy may affect your ability to wear a prosthetic socket, you will be withdrawn from the study if you become pregnant during the course of this study.

A copy of the consent form will be emailed to you at an email address that you provide. It will be a "PDF" document. Most computers already have PDF viewer software installed, which will allow you to open, read, or print the consent form. The email we send you will include a link to PDF viewer software (such as Adobe Acrobat Reader) in case your computer doesn't already have it. If you would prefer to receive a paper copy of the consent form at no cost to you, please contact the researcher listed on page 1 of this consent form.

#### What if I think I have been injured by any research procedures?

If you think you have experienced a medical problem or injury because of participating in this study, please contact Stefania Fatone, PhD, at 206-685-7918 right away. She will refer you for treatment.

The costs of the treatment may be billed to you or your health insurance just like other medical costs, or it may be covered by the UW's discretionary Human Subjects Assistance Program (HSAP), depending on a number of factors. The researcher may request HSAP coverage by following established procedures. If you wish to request HSAP coverage yourself, contact the researcher or the UW Human Subjects Division at <a href="https://hsa.nih.gov/hsa.nih.g

The UW does not normally provide any other form of compensation for injury. However, the law may allow you to seek payment for injury-related expenses if they are caused by malpractice or the fault of the researchers. You do not waive any right to seek payment by signing this consent form.



## **Participant's Statement**

This study has been explained to me. I volunteer to take part in this research. I have had a chance to ask questions. If I have questions later about the research, or if I have been harmed by participating in this study, I can contact one of the researchers listed on the first page of this consent form. If I have questions about my rights as a research subject, I can call the Human Subjects Division at (206) 543-0098. I will receive a copy of this consent form.

Printed name of participant

Signature of participant

Date

## **Consent Presenter Statement**

I have provided this participant and/or their legally authorized representative (LAR) with information about this study. The participant/LAR has been given sufficient time to consider participation and I have answered any questions they had. The participant and/or their LAR indicated that they understand the nature of the study, including risks and benefits of participating.

Printed name of study staff obtaining consent

Date

Copies to:

Researcher Participant